CLINICAL TRIAL: NCT02072837
Title: Dyslipidemia-related Variables as Risk Factor for Cardiovascular Disease in Patients on the End-stage of Renal Disease
Brief Title: Dyslipidemia-related Risk Factors in Dialysis
Status: Completed | Type: Observational
Sponsor: National and Kapodistrian University of Athens (Other)
Responsible Party: Principal Investigator, Vaia D.Raikou, Ph.D Nephrologist; Researcher, National and Kapodistrian University of Athens
Other Study IDs: E.S.931/5-12-2006
Record Dates: First submitted 2014-02-25; First posted 2014-02-27 (Estimated); Last update posted 2014-02-28 (Estimated); Status verified 2014-02

CONDITIONS: Chronic Renal Disease; Cardiovascular Disease; Dyslipidemia
Keywords: hemodialysis, dyslipidemia, cardiovascular disease
MeSH Terms: conditions — Renal Insufficiency, Chronic; Cardiovascular Diseases; Dyslipidemias

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: Yes

SUMMARY:
In this study, we studied lipoprotein abnormalities-related variables as risk factors for the development of cardiovascular disease in patients on renal replacement therapies.We studied 96 dialyzed patients, 62 males and 34 females, on mean age 62.1 years old and 24 healthy controls.We concluded that metabolic acidosis activating the inflammation and lipoprotein oxidation influences the dyslipidemia and cardiovascular morbidity of patients on renal replacement therapies.Dialysis adequacy was positively associated to cardioprotective HDL.Peritoneal dialysis holds a better acidosis level and lower oxidized lipids than hemodialysis modalities.

DETAILED DESCRIPTION:
Blood samples were obtained by venipuncture in the peritoneal dialyzed patients and control group in a twelve hours fasting state.In hemodialyzed patients blood was drawn just before the start of the mean weekly dialysis session also in a twelve hours fasting state from the vascular access.

All samples were received once at baseline time ( in the start of the study ). Peripheral systolic and diastolic blood pressures were calculated as an average of 10 measurements during a renal replacement treatment month in the starting time of the study.

Also, electrocardiographic examination, echocardiography and the calculation of ankle-brachial blood pressure index became once in the start of the study.

ELIGIBILITY:
Inclusion Criteria:

* permanent renal replacement therapy more than 6 months and
* accurate dry body weight

Exclusion Criteria:

* acute illness,
* significant infection,
* malignancy,
* Kt/V for urea <1.2.

Ages: 24 Years to 87 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: We studied 96 dialyzed patients at Nephrology Department of "Laiko, University General Hospital of Athens" and Renal Unit of "Diagnostic and Therapeutic Center of Athens Hygeia SA". 62 males and 34 females participated in this study.The treatment modalities which were applied were : regular haemodialysis (HD, n=34), predilution haemodiafiltration (HDF, n=42) and peritoneal dialysis (PD, n=20).
Sampling Method: Non-Probability Sample
Enrollment: 96 (Actual)
Dates: Start 2012-01; Primary Completion 2014-01 (Actual); Study Completion 2014-01 (Actual)

PRIMARY OUTCOMES:
Associations between dyslipidemia with cardiovascular disease on patients on renal replacement therapy | February 2014

CONTACTS AND LOCATIONS:
Overall Officials: Vaia D. Raikou, Ph.D, Principal Investigator — National & Kapodistrian University of Athens, School of Medicine